CLINICAL TRIAL: NCT00968903
Title: Effects of Pre-operative Methylprednisolone (125mg iv) After Total Hip Arthroplasty: A Prospective, Randomized, Double-blind, Placebo-controlled Trail
Brief Title: Effects of Methylprednisolone After Total Hip Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Lundbeck Foundation (Other)
Responsible Party: Principal Investigator, Troels Haxholdt Lunn, MD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: H-A-2008-030; 2009-41-3784; 2612-3916; EudraCT: 2008-006528-67
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Last update posted 2011-09-29 (Estimated); Status verified 2011-09

CONDITIONS: LOS; Postoperative Pain; Postoperative Nausea and Vomiting; Sleeping Quality; Fatigue; Inflammatory Response
Keywords: Hip arthroplasty; Methylprednisolone; Post-operative pain
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting; Fatigue | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methylprednisolone (Active Comparator): Methylprednisolone 125 mg iv pre-operatively
  Interventions: Drug: Methylprednisolone
- Saline (Placebo Comparator): Saline iv pre-operatively in equivalent volume (placebo)
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Methylprednisolone — Methylprednisolone 125 mg iv pre-operatively

SUMMARY:
The purpose of the study is to compare the effects of pre-operative methylprednisolone (125mg iv) versus placebo on postoperative outcome after hip arthroplasty.

The hypothesis is that pre-operative methylprednisolone (125mg iv) will reduce time to fulfill discharge criteria.

DETAILED DESCRIPTION:
In spite of being one of the last century's most successful surgical procedures in treatment of advanced osteoarthritis total hip arthroplasty is still associated with postoperative pain and delayed rehabilitation. The investigators therefore decided to evaluate the effects of pre-operative methylprednisolone (125mg iv) versus placebo on postoperative outcome in a well defined fast-track setup after hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Elective total hip arthroplasty
* Able to speak and understand danish
* Able to give informed consent

Exclusion Criteria:

* Alcohol or medical abuse
* Allergies to local anesthetics or methylprednisolone
* Age < 18 years
* Daily use of opioids or glucocorticoids
* Pregnancy or breastfeeding (fertile women)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-04; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Time to fulfill discharge criteria | At discharge (mean 1-2 days)

SECONDARY OUTCOMES:
Hand muscle strength | 24 hours
Sleeping quality on the visual analog scale | up to four days
Inflammatory response measured as CRP in blood sample | 24 hours postoperatively
Fatigue measured on a 10 point numeric range scale | up to four days
Additional analgetics, antinausea agents and sleeping medicine. | up to four days
  Measures as mg (analgetics) and daily use (yes or no)(antinausea agents and sleeping medicine).
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | up to 30 days
Postoperative pain scores on the visual analog scale | up 30 days
Postoperative nausea and vomiting (PONV) on 4 point numeric range scale | up to 4 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre University Hospital, Copenhagen, Hvidovre, Denmark